CLINICAL TRIAL: NCT05935553
Title: Baclofen for Improving Benzodiazepine Titration in Benzodiazepine Dependence
Acronym: BABET
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL21_1318; 2022-502307-30-00 (EU CTIS Number)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Benzodiazepine Dependence
Keywords: Benzodiazepine Dependence; baclofen; efficacy
MeSH Terms: interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baclofen 30 microgram (mg) treatment (Experimental): baclofen treatment (30 mg/per day)
  Interventions: Drug: Baclofen 30 mg
- Baclofen 60 mg (Experimental): baclofen treatment (60 mg/per day)
  Interventions: Drug: Baclofen 60 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen 30 mg — * baclofen 10 mg capsule (for the 30 mg-baclofen 30 mg arm)
  * Dosage: 3 capsules of baclofen 10 mg per day
  * route of administration: Oral
  * duration of treatment: Total duration of treatment is 13 weeks including 1 week of dose escalation, 11 weeks of maintenance at full dose, and 1 week of dose de-escalation
  Arms: Baclofen 30 microgram (mg) treatment
Drug: Baclofen 60 mg — * baclofen 20 mg capsule (for the 60 mg baclofen arm)
  * Dosage: 3 capsules of baclofen 20 mg per day
  * route of administration: Oral
  * duration of treatment: Total duration of treatment is 13 weeks including 1 week of dose escalation, 11 weeks of maintenance at full dose, and 1 week of dose de-escalation
  Arms: Baclofen 60 mg
Drug: Placebo — * placebo capsule (for the placebo arm)
  * Dosage:3 capsules of placebo per day
  * route of administration: Oral
  * duration of treatment: Total duration of treatment is 13 weeks including 1 week of dose escalation, 11 weeks of maintenance at full dose, and 1 week of dose de-escalation
  Arms: Placebo

SUMMARY:
Benzodiazepines and related molecules are among the most prescribed psychotropic treatments in France and Europe. 13.4% of the French population had at least one reimbursement of benzodiazepines in 2015, which places France second in Europe.

However, the chronic use of benzodiazepines is a source of numerous complications, particularly addictive. To date, there is no authorized pharmacological treatment for benzodiazepine withdrawal.

Baclofen is a gamma-aminobutyric acid (GABA)-B agonist, a pharmacological receptor that regulates GABA-A, the target of benzodiazepines. The pharmacological mechanisms of baclofen are therefore related to those of benzodiazepines. Empirical use outside of the MA has shown that baclofen can facilitate the reduction of benzodiazepines in cases of severe addiction, but this pharmaceutical interest remains to be demonstrated in a comparative study.

The main objective of the project is to evaluate the efficacy of baclofen, compared to placebo, in reducing benzodiazepine doses in patients with benzodiazepine use disorder (BUD).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years to ≤ 65 years
* For women of childbearing potential :

  * negative pregnancy test at inclusion
  * and use of effective contraception which will be continued throughout the trial period
  * and agrees to carry out pregnancy tests throughout the trial period.
* BUD of any severity defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 criteria
* Average daily benzodiazepine dosage between 50 mg and 200 mg-diazepam (according to Ashton equivalence table) over the 28 days prior to inclusion. Benzodiazepine equivalents (zolpidem, zopiclone and eszopiclone) will be counted as part of the total equivalent daily dose of diazepam and will also be included in the tapering procedure.
* Continued use of benzodiazepines for more than 12 weeks
* At least one history of BUD treatment failure. A treatment failure is defined as a failure to withdraw from the full dose (i.e., discontinuation of benzodiazepine and related prescriptions) according to a previously established tapering schedule, by a general practitioner or specialist
* Patient affiliated to a social security system.
* Patients with or without guardianship
* Patient capable of giving free, informed and written consent.

Exclusion Criteria:

* Cirrhosis of the liver
* Patients with significant medical conditions such as cancer, HIV, epilepsy, chronic respiratory failure, renal failure, etc.
* Non-compatible health conditions (at the discretion of the investigator)
* The following psychiatric conditions as defined by DSM-5 criteria: schizophrenic disorder, persistent delusional disorder, schizophreniform disorder, schizoaffective disorder, bipolar disorder, autism spectrum disorder identified using the Mini International Neuropsychiatric Interview version 7.0.2 (MINI 7.0.2)
* Suicidal state identified using MINI 7.0.2
* Dependence on substances or drugs other than benzodiazepines and nicotine (dependence will be identified through the use of MINI 7.0.2)
* History of baclofen use for all indications
* Unauthorized combination therapies will be: pregabalin, topiramate, ketamine, sodium oxybate, gabapentin, valproic acid, sodium valproate, melatonin, buspirone, hydroxyzine, propranolol, bisoprolol, etifoxin, carbamazepine, clonidine, paroxetine, all neuroleptic/antipsychotic class therapies, and tricyclic antidepressants
* Pregnant or nursing women
* Hypersensitivity to baclofen or microcrystalline cellulose.
* Participants under guardianship
* Patients who need to drive and/or use machines during the 1-week dose escalation phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Difference in total benzodiazepine consumption, in mg-diazepam | between the 28 days before inclusion in the clinical trial and the last 28 days of the clinical trial
  This difference will be compared between the two groups (winning baclofen group and placebo group). Total benzodiazepine consumption will be measured using the Benzodiazepine Timeline Follow-Back (B-TLFB). A mean value (in mg/d) for the 28 days of consumption will be calculated for each patient (between the 28 days prior to inclusion in the clinical trial and the last 28 days of the clinical trial).

SECONDARY OUTCOMES:
Frequency of serious adverse events of special interest | through study completion, an average of 4 and a half months
  The frequency of serious adverse events of particular interest will be collected from inclusion to the end of the study for each patient.
Frequency of non-serious adverse events of special interest | through study completion, an average of 4 and a half months
  The frequency of non-serious adverse events of particular interest will be collected from inclusion to the end of the study for each patient.
frequency of all-cause study discontinuations | through study completion, an average of 4 and a half months
  frequency of all-cause study discontinuations will be collected from inclusion to the end of the study for each patient.
Frequency of benzodiazepine discontinuation at the last visit of the treatment period by urine test | at study completion, an average of 4 and a half months
  Toxicology will be measured by a urine test during the last visit of the treatment period.
Frequency of benzodiazepine discontinuation at the last visit of the treatment period by B-TLFB questionnaire | at study completion, an average of 4 and a half months
  Frequency of benzodiazepine discontinuation at the last visit of the treatment period will collected by B-TLFB questionnaire.
  The B-TLFB involves asking patients to retrospectively estimate their benzodiazepine consumption.
Frequency of benzodiazepine discontinuation at the last visit of the treatment period by the Clinical Institute Withdrawal Assessment of Benzodiazepine (CIWA-B) questionnaire | up to visit 6, an average of 3 and a half months
  The severity score for benzodiazepine withdrawal will be assessed at visit 1 to visit 6 by the Clinical Institute Withdrawal Assessment of Benzodiazepine (CIWA-B).The B-TLFB involves asking patients to retrospectively estimate their benzodiazepine consumption.
  The CIWA-B comprises client-reported symptoms and clinical observations. Questions 1-11 and 13-17 are client-reported symptoms, with each scored on five-point scales from 0 = not at all to 4 = very much so. Question 12 is also a client-reported item, but the 5 scale is reversed, i.e., 0 = Very much so to 4 = Not at all. Questions 18-20 are clinical observations, with all three scored on five-point scales (i.e. 0, 1, 2, 3 or 4).
  A total score is obtained by summing questions 1-20: The minimum total score possible is 0, and the maximum total score possible is 80.
  1-20 Mild withdrawal 21-40 Moderate withdrawal 41-60 Severe withdrawal 61-80 Very severe withdrawal
Craving score assessed by the Visual Analog Scale (VAS) | up to visit 6, an average of 3 and a half months
  Craving score assessed by the Visual Analog Scale (VAS) will be collected at visit 1 to visit 6.
Anxiety symptoms assessed by the State Trait Inventory Anxiety (STAI-Y) | up to visit 6, an average of 3 and a half months
  Anxiety symptoms will be evaluated by the State Trait Inventory Anxiety (STAI-Y) collected at visit 1 and visit 6. It is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Higher scores are positively correlated with higher levels of anxiety. Its most current revision is Form Y and it is offered in more than 40 languages.
Depression score assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) | up to visit 6, an average of 3 and a half months
  Depression score will be evaluated by the MADRS questionnaire collected at visit 1 and visit 6.
  It assesses the severity of symptoms in a wide range of areas, such as mood, sleep and appetite, physical and mental fatigue and thoughts of suicide.
  The scale comprises 10 items rated from 0 to 6. 0 to 6 points: the patient is considered to be healthy. 7 to 19 points: the patient is considered to be mildly depressed. 20 to 34 points: the patient is considered to have moderate depression. > 34 points: the patient is considered to have severe depression.
Subjective sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI) | up to visit 6, an average of 3 and a half months
  Subjective sleep quality will be evaluated by the PSQI questionnaire collected at visit 1 to visit 6.* The PSQI consists of 19 self-assessment questions and 5 questions asked of the spouse or roommate (if any). Only the self-assessment questions are included in the score.
  The 19 self-assessment questions combine to give 7 'components' of the overall score, with each component receiving a score from 0 to 3.
  In all cases, a score of 0 indicates that there are no difficulties, while a score of 3 indicates the existence of severe difficulties. The 7 components of the score are added together to give an overall score ranging from 0 to 21 points, with 0 meaning that there are no difficulties, and 21 indicating major difficulties.
Quality of life (SF-12 v2) | up to visit 6, an average of 3 and a half months
  The SF-12 questionnaire will be collected to visit 1 and visit 6. It is a 12-item short-form health survey that assesses the same eight health domains as the SF-36v2® Health Survey, acting as an abridged version with one or two questions per domain: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Lower scores indicating better physical and mental health functioning

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier le Vinatier, Bron
  - Hôpital Edouard Herriot, Lyon